CLINICAL TRIAL: NCT00141830
Title: A Randomized, Parallel, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of 3 Oral Doses of ERB-041 in Subjects With Rheumatoid Arthritis on a Background of Methotrexate Therapy
Brief Title: Study Evaluating ERB-041 With Methotrexate in Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3142A1-202; B2381010 (Other: Pfizer); 2005-001319-23 (EudraCT Number)
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; ERB 041

INTERVENTIONS:
Drug: Methotrexate plus ERB-041 for 12 weeks
Drug: Placebo for 12 weeks

SUMMARY:
The primary objective of this study is to compare the efficacy and safety of 3 dose levels of oral ERB-041 administered daily for 12 weeks versus placebo in subjects with active rheumatoid arthritis who have had a suboptimal response to therapy with stable doses of methotrexate (MTX).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of active rheumatoid arthritis for at least 6 months and on a stable dose of methotrexate for at least 12 weeks
* Rheumatoid arthritis onset after 16 years of age

Exclusion Criteria:

* Any significant health problem other than rheumatoid arthritis
* History of male or female reproductive system cancer
* Clinically significant laboratory abnormalities

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2005-08; Primary Completion 2006-10-19 (Actual); Study Completion 2006-10-19 (Actual)

PRIMARY OUTCOMES:
-ACR 20 response at Week 12

SECONDARY OUTCOMES:
Secondary efficacy measures include ACR 50 and ACR 70 response.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For South Africa, please contact ZAFinfo@wyeth.com
Locations (35):
- United States (14):
  - Largo, Florida
  - Palm Harbor, Florida
  - Sarasota, Florida
  - Boise, Idaho
  - Kansas City, Kansas
  - Frederick, Maryland
  - Albuquerque, New Mexico
  - Charlotte, North Carolina
  - Duncansville, Pennsylvania
  - Austin, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Spokane, Washington
  - La Crosse, Wisconsin
- Canada (7):
  - Penticton, British Columbia
  - Newmarket, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Trois-Rivières, Quebec
  - Saskatoon, Saskatchewan
  - Québec
- Hungary (3):
  - Békéscsaba
  - Budapest
  - Veszprém
- Italy (5):
  - Brescia
  - Genova
  - Pavia
  - Roma
  - Siena
- Mexico (2):
  - Jalisco, Guadalajara
  - Delegacion Cuahutemoc
- Spain (4):
  - Andalucia, Andalusia
  - Castilla La Mancha
  - Comunidad Valenciana
  - Madrid

REFERENCES:
- [Derived] Roman-Blas JA, Castaneda S, Cutolo M, Herrero-Beaumont G. Efficacy and safety of a selective estrogen receptor beta agonist, ERB-041, in patients with rheumatoid arthritis: a 12-week, randomized, placebo-controlled, phase II study. Arthritis Care Res (Hoboken). 2010 Nov;62(11):1588-93. doi: 10.1002/acr.20275. Epub 2010 Jun 15. PMID 20556817